CLINICAL TRIAL: NCT03015792
Title: Phase I/II Trial of Ibrutinib, Dexamethasone, and Lenalidomide as Initial Therapy for Transplant Ineligible Multiple Myeloma Patients
Brief Title: Ibrutinib, Lenalidomide, and Dexamethasone in Treating Patients With Multiple Myeloma Ineligible for Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug company decided to not fund the phase 2 portion
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC148A; NCI-2017-00006 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ibrutinib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, lenalidomide, dexamethasone) (Experimental): PHASE I: Patients receive ibrutinib PO on days 1-28, lenalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Beginning course 25, patients receive lenalidomide PO on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 84 days in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive ibrutinib and dexamethasone as in phase I and lenalidomide PO on days 1-21 beginning course 2. Beginning course 25, patients receive lenalidomide and dexamethasone as in phase I.
  Interventions: Drug: Dexamethasone; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Pharmacological Study; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase I/II trial studies the best dose and side effects of ibrutinib when given together with lenalidomide and dexamethasone and how well they work in treating patients with multiple myeloma that are not eligible for transplant. Ibrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as lenalidomide and dexamethasone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ibrutinib, lenalidomide, and dexamethasone may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of ibrutinib that can be combined with lenalidomide and dexamethasone in relapsed multiple myeloma (MM) patients. (Phase I) II. To estimate the overall response rate (ORR) including partial response (PR) or better of the combination of ibrutinib, lenalidomide, and dexamethasone in subjects with newly diagnosed MM who are not candidates for high dose chemotherapy and autologous stem cell transplantation (ASCT). (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of this regimen in relapsed MM patients. (Phase I) II. To evaluate the progression free survival (PFS) of the combination of ibrutinib, lenalidomide, and dexamethasone in MM patients. (Phase II) III. To evaluate the safety profile of this regimen in untreated MM patients. (Phase II) IV. To evaluate the duration of response for patients treated with this 3-drug regimen. (Phase II) V. To evaluate overall survival (OS) for patients treated with this 3-drug regimen. (Phase II)

EXPLORATORY OBJECTIVES:

I. To explore compliance to treatment. II. To assess effects of treatment on patient-reported quality of life (QoL) measures.

CORRELATIVE RESEARCH OBJECTIVES:

I. To determine the role of members of the BTK signalosome in achievement or lack thereof of response to ibrutinib.

II. To explore biologic effects of ibrutinib on microenvironment in MM and correlate with response to treatment.

III. To evaluate pharmacodynamic measures including receptor occupancy for BTK prior to introducing lenalidomide in patients treated with ibrutinib and dexamethasone.

IV. To evaluate the impact of ibrutinib on platelet aggregation.

OUTLINE: This is a phase I, dose-escalation study of ibrutinib followed by a phase II study.

PHASE I: Patients receive ibrutinib orally (PO) on days 1-28, lenalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Beginning course 25, patients receive lenalidomide PO on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 84 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients receive ibrutinib and dexamethasone as in phase I and lenalidomide PO on days 1-21 beginning course 2. Beginning course 25, patients receive lenalidomide and dexamethasone as in phase I.

After completion of study treatment, patients are followed up every 3 months, then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis

  * Phase I: confirmed diagnosis of relapsed or refractory multiple myeloma
  * Phase II: confirmed diagnosis of active multiple myeloma and must be newly diagnosed
  * NOTE: all tests for establishing disease status must be completed =< 28 days prior to registration
* Measurable disease =< 28 days prior to registration, defined by at least one of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * > 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * Serum immunoglobulin free light chain > 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis > 30% (evaluable disease)
* Prior treatment

  * Phase I: exposure to 2-3 prior lines of therapy or no therapeutic options
  * Phase II: previously untreated for symptomatic MM
  * EXCEPTION: =< 7 days with pulse steroids or localized radiation therapy, without curative intent, for a myeloma-related complication prior to registration is allowed, as considered necessary by the treating physician
* Myeloma Frailty Score:

  * NOTE: this will include calculating a frailty score (based on age, activities of daily living, instrumental activities of daily living and Charlson comorbidity index)

    * Phase I: "intermediate fitness" or "frail"; NOTE: no "fit" patients will be included in the phase 1 portion of the trial which is being done to determine the MTD of the 3-drug combination
    * Phase II: transplant-ineligible as per their treating physician; NOTE: all the patients with "intermediate fitness" or "frail" status will be considered transplant-ineligible; other reasons to consider transplant ineligibility may include, but are not limited to: financial constraints or patient preference; in case such patients have a frailty score of "fit", it should be duly noted by the treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,000 cell/mm^3 without growth factor support (obtained =< 14 days prior to registration)
* Platelets >= 50,000 cells/mm^3 for patients who have bone marrow (obtained =< 14 days prior to registration)
* Plasmacytosis < 50% or >= 30,000 cells/mm^3 for patients who have bone marrow plasmacytosis of >= 50% (obtained =< 14 days prior to registration)
* Calculated or measured creatinine clearance >= 30 ml/min (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilbert's syndrome (obtained =< 14 days prior to registration)
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 3 x ULN (obtained =< 14 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5 X ULN (obtained =< 14 days prior to registration)
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Persons able to become pregnant must be willing to adhere to the scheduled pregnancy testing as required in the REVLIMID Risk Evaluation and Mitigation Strategy (REMS) program
* Willing to be registered into the mandatory REVLIMID REMS program, and willing and able to comply with the requirements of the REVLIMID REMS program
* Ability to complete study-related (QoL, pill diary) questionnaire(s) by themselves or with assistance
* Willing to provide bone marrow aspirate and core, and blood samples for correlative research purposes

Exclusion Criteria:

* Non-secretory MM or known amyloid light-chain (AL) amyloidosis
* Clinically significant active infection requiring intravenous antibiotics =< 14 days prior to registration
* >= grade 3 neuropathy and/or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Other prior malignancy; EXCEPTIONS:

  * Adequately treated basal cell or squamous cell skin cancer
  * Any in situ cancer
  * Adequately treated stage I or II cancer from which the patient is currently in complete remission, or
  * Any other cancer from which the patient has been disease-free for >= at least three years prior to registration
* Concurrent therapy considered to be investigational; NOTE: patients must not be planning to receive any radiation therapy (except localized radiation for palliative care that must be completed prior to starting cycle 1, day 1)
* Any of the following:

  * Pregnant women
  * Nursing women (lactating females are eligible provided that they agree not to breast feed while taking lenalidomide)
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Requires treatment with a strong cytochrome (CYP) 3A4/5 inhibitor
* Major surgery =< 4 weeks prior to registration
* History of stroke/intracranial hemorrhage =< 6 months prior to registration
* Requires use of therapeutic anticoagulation prior to registration

  * NOTE: thromboprophylaxis with any agent is permitted
* History of clinically significant bleeding or known platelet or coagulation disorder
* Clinically significant cardiac illness including New York Heart Association (NYHA) class III or class IV heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, or >= grade 3 cardiac arrhythmias noted =< 14 days prior to registration
* Hepatic impairment:

  * Phase I: any currently active, clinically significant hepatic impairment (Child-Pugh class A, B, or C according to the Child Pugh classification)
  * Phase II: currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification
* Known human immunodeficiency virus (HIV) positive (+) patients; EXCEPTION: if they meet the following additional criteria =< 28 days prior to registration:

  * CD4 cells >= 500/mm^3
  * Viral load of < 50 copies HIV messenger (m) ribonucleic acid (RNA)/mm^3 if on combination antiretroviral therapy (cART) or < 10,000 copies HIV mRNA if not on cART • No zidovudine or stavudine as part of cART
* Known hepatitis B or hepatitis C infection; EXCEPTION: if viral load < 800,000 IU/L
* Phase I: active dermatologic disease >= grade 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0 (Phase I) | Up to 28 days
Rate of confirmed response defined as patient who has achieved a stringent (s) complete response (CR), CR, very good partial response (VGPR), or partial response (PR) on two consecutive evaluations at any time during treatment (Phase II) | Up to 3 years
  Response will be evaluated using all cycles of treatment. Responses will be summarized by simple descriptive summary statistics delineating depth of response as well as stable and progressive disease in this patient population. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Progression-free survival (Phase II) | From registration to the time of progression or death due to any cause, assessed up to 3 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Overall survival (Phase II) | From registration to death due to any cause, assessed up to 3 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Duration of response (Phase II) | The date at which the patient's objective status is first noted to be a sCR, CR, VGPR, or PR to the earliest date progression is documented, assessed up to 3 years
  The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Incidence of adverse events assessed by CTCAE v 4.0 (Phase II) | Up to 30 days after last dose of study treatment
  The number and severity of all adverse events (overall and by dose-level) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion. Overall toxicity incidence as well as toxicity profiles by dose level and patient will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.

OTHER OUTCOMES:
Compliance to treatment (Phase II) | Up to 3 years
  Patient compliance to ibrutinib, dexamethasone, and lenalidomide will be assessed by means of self-reported and healthcare staff assessed pill count/diary. Correlation between medication adherence and disease response will be assessed.
QoL measured by the MD Anderson Symptom Inventory - Multiple Myeloma (Phase II) | Up to 3 years
BTK signalosome members (Phase II) | Up to 3 years
  Will be profiled by MSD-based mesoscale assay (or phospho-flow) at baseline before treatment, after cycle 1 (phase II patients only), and at the time of response assessment or disease progression. BTK signalosome component expression levels will be determined from BM and/or peripheral blood. Each measure will be summarized descriptively at each time point and changes across time will be evaluated. Correlation with response to overall therapy will be assessed using Wilcoxon's rank sum tests.
T-cells populations modulation (Phase II) | Up to 3 years
  Will conduct flow cytometry/fluorescence activated cell sorting (FACS) analysis to identify percentages of the immune cell populations (T-cells, natural killer cells, macrophages) in the bone marrow and peripheral blood at baseline before treatment, after cycle 1 (phase II patients only) and at the time of response assessment or disease progression. Each measure will be summarized descriptively at each time point and changes across time will be evaluated. Correlation with response to overall therapy will be assessed using Wilcoxon's rank sum tests.

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Ailawadhi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT03015792/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT03015792/ICF_001.pdf